CLINICAL TRIAL: NCT01424202
Title: Effects of Mechanical Insufflation-Exsufflation in Preventing Respiratory Failure After Extubation
Acronym: MIEICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Miguel R. Goncalves, Professor, Hospital Sao Joao
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MIEICU-08112010
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Post-extubation Failure; Persistent Weaning Failure; Secretion Encumbrance; Weak Cough; Ventilatory Failure
Keywords: Post extubation failure; Mechanical Insufflation-Exsufflation; Noninvasive Ventilation; Weaning
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B (Experimental): Patients received (post-extubation) standard medical treatment (SMT), including NIV in case of specific indications plus daily sessions of mechanical in-exsufflation (MI-E).
  Interventions: Device: Mechanical Insufflation Exsufflation
- Group A (No Intervention): Patients received (post-extubation) standard medical treatment (SMT), including NIV in case of specific indications.

INTERVENTIONS:
Device: Mechanical Insufflation Exsufflation — After passing the SBT and randomized to group B, before extubation, all patients were submitted to a treatment of MI-E (3 sessions) through the endotracheal tube with pressures set at 40 cm H2O for insufflation and -40 cm H2O for exsufflation pressure. An insufflation/exsufflation time ratio of 3secs/2 secs and a pause of 3 sec between each cycle was used. Eight cycles were applied in every session with an abdominal thrust timed to the exsufflation cycle.
  On top of the standard medical therapy, during the first 48 hours post extubation, each patient received 3 daily treatments by means of a light-weight, elastic oronasal mask. Treatments (3 sessions each) were divided between morning, afternoon and night, making a total of 9 daily sessions.
  The daily treatment frequency and its outcomes were recorded in a diary by the nursing staff. All MI-E treatments were administered by a trained respiratory therapist, ICU physician or nurse.
  Arms: Group B

SUMMARY:
Weaning protocols that include the use of noninvasive ventilation (NIV), decreases the incidence of re-intubation and ICU length of stay. However, the role of NIV in post-extubation failure is still not clear. Impaired airway clearance is associated with NIV failure. Mechanical Insufflation-Exsufflation (MI-E) is an assisted coughing technique that has been proven to be very effective in patients under NIV.

In this study the investigators assess the efficacy of MI-E as part of a protocol for patients that develop respiratory failure after extubation.

DETAILED DESCRIPTION:
Patients under mechanical ventilation (MV) for more than 48 hours with specific inclusion criteria, who successfully tolerated an spontaneous breathing trial (SBT) were randomly allocated before extubation, either for (A) conventional extubation protocol (control group) or (B) MI-E extubation protocol (study group). Re-intubation rates, ICU length of stay and NIV failure rates were analyzed.

Inclusion of MI-E in post-extubation failure may reduce re-intubation rates with consequent reduction in post-extubation ICU length of stay. This technique seems to be efficient in improving the efficacy of NIV in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and under mechanical ventilation, for more than 48 hours, for acute hypoxemic and/or hypercapnic respiratory failure from a specific etiology

Exclusion Criteria:

* facial or cranial trauma, tracheostomy, active upper gastrointestinal bleeding, neurologic instability (inability to respond to direct simple orders), hemodynamic instability, lack of cooperation and confirmed diagnosis of neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
re-intubation rates | 48 hours

SECONDARY OUTCOMES:
NIV failure rates | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care and Emergency Department;, Faculty of Medicine, University Hospital of S. João, Porto, Porto District, Portugal

REFERENCES:
- [Result] Esteban A, Frutos-Vivar F, Ferguson ND, Arabi Y, Apezteguia C, Gonzalez M, Epstein SK, Hill NS, Nava S, Soares MA, D'Empaire G, Alia I, Anzueto A. Noninvasive positive-pressure ventilation for respiratory failure after extubation. N Engl J Med. 2004 Jun 10;350(24):2452-60. doi: 10.1056/NEJMoa032736. PMID 15190137